CLINICAL TRIAL: NCT01697215
Title: Novel Device (AirWave™) to Assess Endotracheal Tube Migration.
Brief Title: Novel Device to Assess Endotracheal Tube Migration
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Adriano Tonelli, Staff Physician, The Cleveland Clinic
Other Study IDs: 111128-PIP
Record Dates: First submitted 2012-09-21; First posted 2012-10-02 (Estimated); Results first posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Mechanically Ventilated Patients Admitted to a MICU

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Oral or nasal endotracheal intubation: Oral or nasal endotracheal intubation, anticipated to last at least 48 hours Adults that require ETT internal diameter sizes of 6.5 - 9.0 mm Subject must be at least 18 years old (no upper age limitation) English speaking patients/decision makers.
  Interventions: Other: AirWave

INTERVENTIONS:
Other: AirWave

SUMMARY:
To evaluate the ability of the SonarMed AirWave to provide clinicians with information that enables them to confirm continuous proper placement of the endotracheal tube. This initial study is prospective, observational, looking at CXR results, and comparing those to AirWave system output data.

ELIGIBILITY:
Inclusion Criteria

Subjects will be eligible for inclusion in the study if they meet ALL of the following criteria:

* Oral or nasal endotracheal intubation, anticipated to last at least 48 hours
* Adults that require ETT internal diameter sizes of 6.5 - 9.0 mm
* Subject must be at least 18 years old (no upper age limitation)
* English speaking patients/decision makers.

Exclusion Criteria

* Subjects ventilated through a tracheostomy
* Subjects under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MICU Based
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2012-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adriano Tonelli, MD, Principal Investigator — The Cleveland Clinic Foundatin
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During the study period, 42 patients were enrolled. Subjects had the AirWave system placed within 24 hours of endotracheal intubation. A total of 19 patients had measurements of ETT migration at 24 hours by the three methodologies used in this study.
Pre-assignment Details: Inclusion Criteria: subjects were eligible for the study if they met all of the following criteria: (1) age > 18 years old; (2) oral endotracheal intubation within 24 hours of recruitment; (3) expected duration of mechanical ventilation > 24 hours; (4) ETT internal diameter sizes from 6.5 to 9.0 mm. Exclusion criteria: subjects were excluded from participation if (1) ventilated through a tracheostomy, (2) unable to obtain consent, or (3) pregnancy.
Groups:
- Oral or Nasal Endotracheal Intubation: Oral or nasal endotracheal intubation, anticipated to last at least 48 hours Adults that require ETT internal diameter sizes of 6.5 - 9.0 mm Subject must be at least 18 years old (no upper age limitation) English speaking patients/decision makers.
  AirWave
  Migration at 24 hours as determined by (a) portable CXR (n = 28) was -0.06 (±1.3) cm with range of -3.5 and +3 cm, (b) ETT distance at the lips (n = 38) was -0.29 (±0.93) with a range of -2 to +3, and (c) the AirWave system (n = 27) was 0.39 (±1.5) with a range of -3 to +4 cm. Diverse reasons (Fig. 2) reduced the total number of patients in whom these three techniques can be compared.
Period: Overall Study
Arm/Group | Oral or Nasal Endotracheal Intubation
Started | 42
Migration at 24 hs by CXR | 28
ETT Distance at the Lips | 38
Airwave System | 27
Completed | 19
Not Completed | 23
Not completed — Physician Decision | 5
Not completed — Malfunction | 9
Not completed — CXR not available | 9

BASELINE CHARACTERISTICS:
Groups:
- (ETT) Migration During Routine Care Among Critically Ill Patients: A total of 42 patients (age: 61 [SD ±13] years, men: 52%) were recruited. A total of 19 patients had measurements of ETT migration at 24 hours by the 3 methodologies used in this study.
Arm/Group | (ETT) Migration During Routine Care Among Critically Ill Patients
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 22
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 42

OUTCOME MEASURES:

1. Primary Outcome: Endotracheal Tube Displacement Bias Measured by a Novel Device (AirWave) Compared to CXR
Description: Comparison of migration at 24 hours as measured by the AirWave system and portable CXR using a Bland-Altman analysis.
Time Frame: 24 hours
Population: A total of 19 patients had measurements of ETT migration at 24 hours by the three methodologies used in this study.
Measure: Mean (Standard Deviation); unit: cm
Groups:
- Oral or Nasal Endotracheal Intubation: Oral or nasal endotracheal intubation, anticipated to last at least 48 hours Adults that require ETT internal diameter sizes of 6.5 - 9.0 mm Subject must be at least 18 years old (no upper age limitation) English speaking patients/decision makers.
  AirWave
Arm/Group | Oral or Nasal Endotracheal Intubation
Number analyzed (Participants) | 42
cm
  Migration measured by CXR: number analyzed (Participants) | 28
  Migration measured by CXR | -0.06 (1.3)
  Migration measured by EET lip distance: number analyzed (Participants) | 38
  Migration measured by EET lip distance | -0.29 (0.93)
  Migration measured by AirWave System: number analyzed (Participants) | 27
  Migration measured by AirWave System | 0.39 (1.5)

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Oral or Nasal Endotracheal Intubation
All-Cause Mortality (participants affected / at risk) | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42
Other Adverse Events (participants affected / at risk) | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes